CLINICAL TRIAL: NCT00592683
Title: A Randomized Placebo Controlled Clinical Trial of Omega-3 Fatty Acid Adjunctive to Open-Label Aripiprazole for the Treatment of Bipolar Disorder in Children and Adolescents Ages 6-17 With Bipolar Spectrum Disorder
Brief Title: Omega-3 Fatty Acid Adjunctive to Open-Label Aripiprazole for the Treatment of Bipolar Disorder in Children and Adolescents
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Supply Omega-3 Fatty Acids expired and supplier no longer made same composition.
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Janet Wozniak, MD, Assistant Professor of Psychiatry at Harvard Medical School and at Massachusetts General Hospital, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-P-000413
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Results first posted 2012-04-06 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-03

CONDITIONS: Pediatric Bipolar Disorder
Keywords: bipolar disorder; fish oil; aripiprazole; children
MeSH Terms: conditions — Bipolar Disorder | interventions — Aripiprazole; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aripiprazole plus Fish Oil (Active Comparator): Subjects administered aripiprazole and randomized to receive fish oil
  Interventions: Drug: Aripiprazole; Dietary Supplement: fish oil
- Aripiprazole plus Placebo (Placebo Comparator): Subjects administered aripiprazole and randomized to receive placebo
  Interventions: Drug: Aripiprazole; Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — tablet, start at 2mg and increase/decrease each week, taken daily for 12 weeks
  Other Names: Abilify
Dietary Supplement: fish oil — 1600mg (4 capsules) daily for 12 weeks
  Arms: Aripiprazole plus Fish Oil
Drug: Placebo — Placebo
  Arms: Aripiprazole plus Placebo

SUMMARY:
This will be a 12 week, double blind study of omega-3 fatty acids vs. placebo adjunctive to open-label aripiprazole treatment in children and adolescents (ages 6-17) who meet DSM-IV criteria for bipolar disorder (BPD) (currently manic or mixed). Specific hypotheses are as follows:

Hypothesis 1: Omega-3 fatty acids will be well-tolerated and efficacious in the treatment of children and adolescents with BPD

Hypothesis 2: The total dose of aripiprazole will be lower in those subjects receiving active omega-3 treatment

DETAILED DESCRIPTION:
Initial clinical evidence suggests that the omega-3 fatty acids EPA (eicosapentaenoic acid) and/or DHA (docosahexaenoic acid) may play a therapeutic role in the management of mood disorders. EPA is an essential fatty acid, which can be metabolized to DHA and is a component of the human diet if fish is consumed. Aripiprazole is a novel second general antipsychotic that seems to function as a partial agonist at the dopamine D2 and serotonin 5-HT 1A receptors as well as an antagonist at the serotonin 5-HT 2A receptor. Since it has a favorable adverse event profile in adults, it is an attractive choice for the treatment of youth with bipolar disorder if proven efficacious. Although pilot research showed that omega-3 fatty acids monotherapy treatment resulted in improvement of manic symptoms, the improvement is less dramatic than that observed in trials of antipsychotics. We will test the safety and efficacy of omega-3 fatty acids versus placebo as an adjunctive treatment to open-label aripiprazole in children and adolescents with bipolar disorder.

The proposed study includes 1) the use of a 12-week design to document the response rate 2) careful assessment of safety and tolerability

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject, 6-17 years of age
2. Subject has a DSM-IV diagnosis of bipolar I, bipolar II, or bipolar spectrum disorder and currently displaying manic, hypomanic, or mixed symptoms (with or without psychotic features)
3. Subject and their legal representative have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol
4. Subject and their legal representative must be considered reliable
5. Subject and his/her authorized legal representative must understand the nature of the study. The subject's authorized legal representative must sign an informed consent document and the subject must sign an informed assent document
6. Subject must have an initial score on the Young-Mania Rating Scale (Y-MRS) of at least 20
7. Subject must be able to participate in mandatory blood draws
8. Subject must be able to swallow pills
9. Subjects with comorbid Attention Deficit Hyperactivity Disorder (ADHD), Oppositional Defiant Disorder (ODD), Conduct Disorder (CD), Obsessive Compulsive Disorder (OCD), Pervasive Developmental Disorders (PDD), anxiety and depressive disorders will be allowed to participate in the study provided they do not meet for any of exclusionary criteria
10. For concomitant therapy used to treat ADHD, subject must have been on a stable dose of the medication for 1 month prior to study enrollment. The dose of the ADHD therapy may not change throughout the duration of the study.

Exclusion Criteria:

1. Investigator and his/her immediate family; defined as the investigator's spouse, parent, child, grandparent, or grandchild
2. Serious, unstable illness including heptic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease
3. Uncorrected hypothyroidism or hyperthyroidism
4. History of sensitivity to omega-3 fatty acids. A non-responder or history of intolerance to omega-3 fatty acid, after treatment at adequate doses as determined by the clinician.
5. Severe allergies or multiple adverse drug reactions.
6. Non-febrile seizures without a clear and resolved etiology
7. DSM-IV substance (except nicotine or caffeine) dependence within past 6 months
8. Judged clinically to be at serious suicidal risk
9. Any other concomitant medication with primarily central nervous system activity other than specified in the Concomitant Medication portion of the protocol.
10. Current diagnosis of schizophrenia
11. Pregnant or nursing females

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wozniak, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://massgeneral.org/pediatricpsych/home.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole + Fish Oil: treatment with aripiprazole + fish oil
- Aripiprazole + Placebo: treatment with aripiprazole + placebo
Period: Overall Study
Arm/Group | Aripiprazole + Fish Oil | Aripiprazole + Placebo
Started | 10 | 10
Completed | 6 | 6
Not Completed | 4 | 4
Not completed — Found ineligible | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Study drug expired | 1 | 0
Not completed — Other | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole + Fish Oil | Aripiprazole + Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.8 (3.65) | 11 (3.71) | 10.9 (3.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Bipolar Symptoms as Assessed by Young-Mania Rating Scale (YMRS)
Description: The YMRS is used to evaluate symptoms of mania in children and adolescents. Items are rated from 0-4 or 0-8, with higher scores indicating greater severity. The minimum total score (least severe) is 0, and the maximum total score (most severe) is 60.
Time Frame: weekly for 1st 6 weeks then biweekly
Population: 14 subjects came in for week 12 assessments - included in final analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aripiprazole + Fish Oil | Aripiprazole + Placebo
Number analyzed (Participants) | 8 | 6
Units on a scale | 9.5 (7.78) | 8.5 (7.40)

2. Secondary Outcome: DSM-IV Mania Symptom Checklist
Description: The DSM-IV Mania Symptom Checklist is used to evaluate symptoms of mania. Item scores range from 0-3, with larger scores indicating greater severity. With 33 items, the maximum (most severe) score possible is 99, with the minimum (least severe) score possible being 0.
Time Frame: weekly for first 6 weeks then biweekly
Population: 14 subjects came in for week 12 assessments - included in final analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aripiprazole + Fish Oil | Aripiprazole + Placebo
Number analyzed (Participants) | 8 | 6
units on a scale | 5.25 (5.23) | 5 (3.16)

ADVERSE EVENTS:
Arm/Group | Aripiprazole + Fish Oil | Aripiprazole + Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 9/10 | 9/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole + Fish Oil (N=10) | Aripiprazole + Placebo (N=10)
chest pain with inspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cold symptoms (General disorders) | 0 (0) | 1 (2)
decreased energy (General disorders) | 2 (2) | 1 (1)
decreased appetite (General disorders) | 0 (0) | 2 (3)
diarrhea (Gastrointestinal disorders) | 2 (4) | 0 (0)
dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (3)
dry mouth (General disorders) | 2 (3) | 0 (0)
ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
flatulence (Gastrointestinal disorders) | 1 (2) | 0 (0)
hand tremor (General disorders) | 0 (0) | 1 (1)
headache (General disorders) | 0 (0) | 3 (5)
heartburn (Gastrointestinal disorders) | 0 (0) | 1 (3)
increased appetite (General disorders) | 1 (2) | 2 (2)
increased sleep (General disorders) | 1 (2) | 0 (0)
irritability (General disorders) | 0 (0) | 1 (1)
left ankle swelling (injury) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
period 1 week late (Reproductive system and breast disorders) | 0 (0) | 1 (1)
nausea/vomiting (Gastrointestinal disorders) | 3 (4) | 4 (7)
rash (poison ivy) (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
restless (General disorders) | 0 (0) | 1 (1)
rhinorrhea (General disorders) | 2 (4) | 1 (1)
saddness/crying (Psychiatric disorders) | 0 (0) | 1 (1)
sedation (General disorders) | 2 (3) | 1 (1)
skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
slurred speech (General disorders) | 0 (0) | 1 (1)
sore throat (General disorders) | 1 (2) | 1 (1)
sores in mouth (healed) (General disorders) | 0 (0) | 1 (1)
sprained finger (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
stomachache (Gastrointestinal disorders) | 1 (1) | 1 (1)
tiredness (General disorders) | 7 (16) | 4 (7)
transient facial flushing (General disorders) | 0 (0) | 1 (1)
weight gain (General disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No